CLINICAL TRIAL: NCT03930316
Title: Using a Portable Monitoring Device for Diagnosing Obstructive Sleep Apnea in Patients With Multiple Co-existing Medical Illnesses
Brief Title: Validation of a Portable Sleep Device in Patients With Co-existing Medical Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Associate consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019.025
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: OSA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- observation (Other): validation of observational arm
  Interventions: Device: NOX T3

INTERVENTIONS:
Device: NOX T3 — portable sleep study device

SUMMARY:
The standard sleep study for diagnosing obstructive sleep apnea (OSA) in patients with co-existing illness is by conducting an attended polysomnography (PSG) with more than 7 channels for recording physiological parameters in the sleep center, as recommended by international guidelines. However the guidelines are more than 10 year old without update. With the growing and aging of the population, there is a need to explore if portable monitoring devices could be used in this group of population, so this group of patients can be managed in a timely manner. Portable monitoring devices have been used widely in patients without significant co-existing illness. These devices record at least 4 physiological parameters for diagnosing OSA and can be performed in an unattended setting e.g. at home because of the simplicity. This can shorten the waiting time for making a diagnosis using PSG.

Eighty patients suspected of OSA, with stable co-existing illnesses, will be recruited for the study. Informed consent will be signed before participation. They will be offered a standard attended PSG in the sleep center. A portable monitoring device "Nox T3" will be hooked up to the patients concurrently during the PSG.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suspect of OSA (with or without symptoms) of age between 18 to 80 years old, with or without significant comorbidities.
* Patients consent of concurrent use of both type I and or type III devices at the same time in hospital setting.

Exclusion Criteria:

* Pregnant patients.
* Patients refuse to have both type I and type III devices used concurrently.
* Patients with any co-existing medical illnesses which are unstable. "Unstable" is defined as:
* Any recent hospital admission within 1 month before the schedule of sleep study
* Any recent change of medication within 1 month before the schedule of sleep study
* Any change in patient conditions requiring medical attention within 1 month before the schedule of sleep study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy of the new portable sleep study device with reference to concurrent PSG. | 1 year
  compare the AHI of NOX T3 with reference to PSG

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong